CLINICAL TRIAL: NCT03680534
Title: Three-dimensional Analysis of the Root Canal Preparation With Reciproc Blue, WaveOne Gold and XP EndoShaper
Brief Title: 3D Analysis of Root Canal Conformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institucion Universitaria Colegios de Colombia (Other)
Responsible Party: Principal Investigator, Javier Caviedes-Bucheli, Head and Professor of Postgraduate Endodontics Department, Institucion Universitaria Colegios de Colombia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JCB001
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Endodontic Disease; Root Canal Infection
Keywords: root canal preparation; single-file preparation techniques; 3D reconstruction
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Root Canal Preparation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reciproc Blue (Experimental): Patients in which root canal from a lower premolar was prepared with the Reciproc Blue technique.
  Interventions: Procedure: Root canal preparation
- WaveOne Gold (Experimental): Patients in which root canal from a lower premolar was prepared with the WaveOne Gold technique.
  Interventions: Procedure: Root canal preparation
- XP EndoShaper (Experimental): Patients in which root canal from a lower premolar was prepared with the XP EndoShaper technique.
  Interventions: Procedure: Root canal preparation

INTERVENTIONS:
Procedure: Root canal preparation — Root canals from lower premolars with extraction indicated were prepared previous to being extracted with either the Reciproc Blue, the WaveOne Gold or the XP EndoShaper single-file techniques.
  Other Names: Root canal instrumentation

SUMMARY:
Aim To evaluate in vivo the shaping ability of the canal with 3 different single-file systems: Reciproc Blue, WaveOne Gold and XP Endo-Shaper, using cone beam computed tomography and 3D reconstructions to measure canal volume increase, centering ability of the instruments and canal transportation in human premolars in vivo.

Methodology Thirty human lower premolars were randomly divided into three groups, in which root canals were prepared using one of these single-file systems: Reciproc Blue, WaveOne Gold, and XP EndoShaper. Root canals were scanned before and after root canal preparation by using CBCT and 3D reconstruction was carried out to evaluate canal volume increase, centering ability of the instrument and canal transportation for each group. Statistical analysis was made for each variable to determine statistically significant differences between groups.

ELIGIBILITY:
Inclusion Criteria:

1. 18-30 years old
2. healthy conditions
3. not medicated with any type of drug
4. non-smoking patients
5. lower premolars indicated for extraction due to orthodontic reasons
6. lower premolar with more than one root canal

Exclusion Criteria:

1. Not willing to participate
2. Pregnant women
3. lower premolars with previous root canal therapy
4. lower premolars with

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-11-19 (Actual)

PRIMARY OUTCOMES:
Root canal volume increase in cubic millimetres after root canal preparation by using the volume command in the Rhinoceros 5.0 software | One day
  The total volume of the root canal measured before and after root canal preparation by using the volume command in the Rhinoceros 5.0 software which gives the volume of a solid in cubic millimetres.
Root canal transportation after preparation assessed by superimposing three-dimensional reconstruction images of pre- and post-preparation | One day
  Deviation of the original anatomy of the canal to the mesial or distal wall after root canal preparation evaluated by superimposing three-dimensional reconstruction images of the canal before and after preparation.
Centring ability of the instruments used to prepare the root canal assessed by determining if canal was enlarged equally to each of its walls | One day
  Ability of the instruments used for root canal preparation to equally enlarge all of the canal walls, evaluated by analysing superimposed three-dimensional reconstructed images of before and after root canal preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Caviedes-Bucheli, Principal Investigator — Institucion Universitaria Colegios de Colombia
Locations (1):
- Facultad de Odontologia, Unicoc, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided